CLINICAL TRIAL: NCT01725386
Title: Study on Xeloda® to Document Its Use in Routine Practice in Patients With Metastatic or Advanced Breast Cancer
Brief Title: An Observational Study of Xeloda (Capecitabine) in Participants With Metastatic or Advanced Breast Cancer
Acronym: XEPAD
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML25640
Record Dates: First submitted 2012-11-08; First posted 2012-11-12 (Estimated); Results first posted 2016-08-12 (Estimated); Last update posted 2016-09-28 (Estimated); Status verified 2016-08

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Capecitabine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Monotherapy: Capecitabine as monotherapy according to prescribing information and normal clinical practice.
  Interventions: Drug: Capecitabine
- Combination Therapy: Capecitabine as part of combination therapy according to prescribing information and normal clinical practice.
  Interventions: Drug: Capecitabine

INTERVENTIONS:
Drug: Capecitabine — Oral tablet(s) administered according to prescribing information
  Other Names: XELODA

SUMMARY:
This observational study will evaluate the routine clinical use and the safety and efficacy of capecitabine (Xeloda®) in participants with metastatic or advanced breast cancer. Eligible participants will be followed for up to 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Adult female participants, >/= 18 years of age
* Cytologic/histopathologic confirmed diagnosis of metastatic breast cancer
* Prescribed capecitabine as in routine clinical practice
* Informed consent signed

Exclusion Criteria:

* Participation in any other clinical trial
* History of severe and unexpected reactions to fluoropyrimidine therapy
* Hypersensitivity to capecitabine or to any of the excipients of fluorouracil
* Known dihydropyrimidine dehydrogenase (DPD) deficiency
* Pregnant or lactating women
* Severe leucopenia, neutropenia, or thrombocytopenia
* Severe hepatic impairment
* Severe renal impairment (creatinine clearance below 30 ml/min)
* Treatment with sorivudine or its chemically related analogues, such as brivudine
* Refusal to give consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with metastatic breast cancer initiated on therapy with capecitabine
Sampling Method: Probability Sample
Enrollment: 274 (Actual)
Dates: Start 2011-03; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (10):
- Pakistan (10):
  - Abbottabad
  - Faisalabad
  - Gujranwala
  - Hyderābād
  - Islamabad
  - Karachi
  - Lahore
  - Multan
  - Peshwar
  - Rawalpindi

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 274 participants were enrolled in the study; of these, 23 participants from 3 centers were excluded from the analysis due to study termination at those 3 centers. The remaining 251 participants were eligible for analysis.
Groups:
- Monotherapy: Capecitabine (XELODA®) as monotherapy according to prescribing information and normal clinical practice.
Period: Overall Study
Arm/Group | Monotherapy | Combination Therapy
Started | 188 | 63
Completed | 13 | 17
Not Completed | 175 | 46
Not completed — Death | 84 | 40
Not completed — Lost to Follow-up | 81 | 6
Not completed — Withdrawal by Subject | 10 | 0

BASELINE CHARACTERISTICS:
Population: Participants eligible for analysis (received at least one dose of study medication and for whom data for at least one follow-up variable were available).
Groups:
- Total: Total of all reporting groups
Arm/Group | Monotherapy | Combination Therapy | Total
Number analyzed (Participants) | 188 | 63 | 251
Age, Continuous [Median (Standard Deviation); unit: years] | 47.00 (12.35) | 45.00 (15.19) | 47.00 (12.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 188 | 63 | 251
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percent of Participants With Capecitabine as a First Line, Second Line, or Third Line Therapy
Description: To document use of Capecitabine regimen in the management of participants with metastatic breast cancer, the choice of Capecitabine monotherapy versus combination therapy was summarized according to whether the selection was for the participant's first, second, or third line of treatment.
Time Frame: Up to approximately 4 years
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Monotherapy | Combination Therapy
Number analyzed (Participants) | 188 | 63
percentage of participants
  First Line | 10.6 | 55.6
  Second Line | 71.8 | 41.3
  Third Line | 17.6 | 3.1

2. Primary Outcome: Percentage of Participants Receiving Concomitant Medications During the Study
Description: Percentage of participants receiving concomitant medications during the study along with their prescribed monotherapy or combination therapy were reported.
Time Frame: Up to approximately 4 years
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Monotherapy | Combination Therapy
Number analyzed (Participants) | 188 | 63
percentage of participants | 17.5 | 23.8

3. Secondary Outcome: Percentage of Participants With Relevant Medical History Assessed at Baseline
Description: To document the metastatic breast cancer participant profile, the percentage of participants with relevant medical history as assessed at baseline was summarized.
Time Frame: Day 1
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Monotherapy | Combination Therapy
Number analyzed (Participants) | 188 | 63
percentage of participants
  History of Other Types of Cancer | 0.5 | 1.6
  Family History of Breast Cancer | 9.6 | 12.7
  History of Co-morbidities | 18.1 | 28.6
  Premenopausal Status | 54.8 | 41.3
  Postmenopausal Status | 45.2 | 58.7

4. Secondary Outcome: Percentage of Participants by Histopathology Grade Diagnosis Assessed at Baseline
Description: To document the metastatic breast cancer participant profile, the percentage of participants with histopathology grade diagnosis of moderately differentiated, well differentiated, poorly differentiated/undifferentiated as assessed at baseline was summarized.
Time Frame: Day 1
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Monotherapy | Combination Therapy
Number analyzed (Participants) | 188 | 63
percentage of participants
  Moderately Differentiated | 42.6 | 42.9
  Well Differentiated | 9.0 | 11.1
  Poorly Differentiated/Undifferentiated | 48.4 | 46.0

5. Secondary Outcome: Mean Survival Time
Time Frame: Up to approximately 4 years
Population: as for baseline characteristics
Measure: Mean (95% Confidence Interval); unit: Months
Arm/Group | Monotherapy | Combination Therapy
Number analyzed (Participants) | 188 | 63
Months | 15.493 [14.169 to 16.817] | 15.417 [13.512 to 17.322]
Statistical Analysis 1: Comparison: Monotherapy vs Combination Therapy; Test type: Superiority or Other; p = 0.895, Log Rank (Mantel-Cox)

6. Secondary Outcome: Percentage of Participants With Adverse Events
Time Frame: Up to approximately 4 years
Population: Safety analysis population (participants who received at least one dose of study medication and had at least one post-baseline safety assessment).
Measure: Number; unit: percentage of participants
Arm/Group | Monotherapy | Combination Therapy
Number analyzed (Participants) | 188 | 63
percentage of participants | 45.2 | 66.7

ADVERSE EVENTS:
Time Frame: Up to approximately 4 years
Description: Safety analysis population (participants who received at least one dose of study medication and had at least one post-baseline safety assessment).
Arm/Group | Monotherapy | Combination Therapy
Serious Adverse Events (participants affected / at risk) | 85/188 | 42/63
Other Adverse Events (participants affected / at risk) | 73/188 | 42/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Monotherapy (N=188) | Combination Therapy (N=63)
Anaemia (Blood and lymphatic system disorders) | 1 | 1
Cardiopulmonary Arrest (Cardiac disorders) | 66 | 27
Disease Progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 3
Vomitting (Gastrointestinal disorders) | 0 | 2
Melena (Gastrointestinal disorders) | 1 | 3
Ascites (Gastrointestinal disorders) | 3 | 4
Hematemesis (Gastrointestinal disorders) | 0 | 3
Head Ache (General disorders) | 1 | 0
Body Ache (General disorders) | 1 | 0
Drowsiness (General disorders) | 1 | 0
High grade fever (General disorders) | 1 | 1
Fever (General disorders) | 0 | 1
Diabetic Coma (General disorders) | 1 | 0
Semi conscous/Unconsciousness (General disorders) | 0 | 3
Multiple Organ Failure (General disorders) | 0 | 1
Hepatorenal failure (Hepatobiliary disorders) | 1 | 0
Hepatic Encephalopathy (Hepatobiliary disorders) | 1 | 1
Hepatic failure with Ascites (Hepatobiliary disorders) | 1 | 0
Fracture (Injury, poisoning and procedural complications) | 1 | 0
Cerebral Inflammation (Infections and infestations) | 1 | 0
Pyogenic Meningitis (Infections and infestations) | 0 | 1
Septicemia & Anaemia (Infections and infestations) | 1 | 0
Infected chest wound (Infections and infestations) | 0 | 1
Jaundice (Investigations) | 4 | 2
Pain in sternum (Musculoskeletal and connective tissue disorders) | 1 | 0
Hemiplegia (Nervous system disorders) | 0 | 1
Generalized Fits (Nervous system disorders) | 2 | 2
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Excessive bleeding from Right breast mass (Reproductive system and breast disorders) | 1 | 0
Nodules on Right chest & Axilla (Reproductive system and breast disorders) | 0 | 1
Acute Renal Failure (Renal and urinary disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 5 | 3
Respiratory Distress/Failure (Respiratory, thoracic and mediastinal disorders) | 10 | 7
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Aspiration Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chest Infection (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Skin cutaneous Infiltration (Skin and subcutaneous tissue disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Monotherapy (N=188) | Combination Therapy (N=63)
Anaemia (Blood and lymphatic system disorders) | 0 | 6
Diarrhea (Gastrointestinal disorders) | 13 | 12
Nausea (Gastrointestinal disorders) | 8 | 13
Stomatitis (Gastrointestinal disorders) | 4 | 13
Vomiting (Gastrointestinal disorders) | 16 | 16
Fatigue (General disorders) | 13 | 6
Peripheral edema (General disorders) | 0 | 6
Pyrexia (General disorders) | 5 | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 6
Bone Pain (Musculoskeletal and connective tissue disorders) | 11 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 8
Hand-and-Foot Syndrome (Skin and subcutaneous tissue disorders) | 20 | 17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.